CLINICAL TRIAL: NCT01792596
Title: Satiety Effects of Protein and Fiber Added to Pasta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 1212E25704
Record Dates: First submitted 2013-01-22; First posted 2013-02-15 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences | interventions — Proteins; Dietary Fiber

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- pasta (Other): 1. Plain pasta
  Interventions: Other: Pasta
- pasta with protein (Other): Pasta with protein
  Interventions: Other: Pasta with protein
- pasta with fiber (Other): Pasta with Fiber
  Interventions: Other: Pasta with Fiber

INTERVENTIONS:
Other: Pasta with protein — Pasta with Protein
  Arms: pasta with protein
Other: Pasta with Fiber — Pasta with Fiber
  Arms: pasta with fiber
Other: Pasta — Pasta
  Arms: pasta

SUMMARY:
The combination of fiber and protein added to pasta will enhance satiety.

DETAILED DESCRIPTION:
Subjects will consume 3 different pasta lunches and satiety will be measured by visual analogue scales. They will consume an ad lib snack after 3 hours and food intake will be measured.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* nonsmoking
* body mass index from 19 - 29

Exclusion Criteria:

* Antibiotic use
* any disease
* weight loss
* food allergies
* high fiber intake
* restrained eater

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
satiety | 180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Slavin, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Department of Food Science and Nutrition, Saint Paul, Minnesota, United States